CLINICAL TRIAL: NCT04703738
Title: A Prospective, Randomized and Controlled Multi-center Study of Geistlich Fibro-Gide® Compared With Connective Tissue Graft for Soft Tissue Volume Augmentation Around Dental Implants
Brief Title: Evaluation of Geistlich Fibro-Gide® in Comparison to CTG for the Treatment Around Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Geistlich Pharma AG (Industry)
Collaborators: Medelis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10808-122
Record Dates: First submitted 2020-11-23; First posted 2021-01-11 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-05

CONDITIONS: Soft Tissue Defect
Keywords: soft tissue augmentation; soft tissue volume; Fibro-Gide; CTG; Geistlich

STUDY DESIGN:
Intervention Model Description: parallel, randomized, controlled, single-blind, multi-centre clinical trial
Who Masked: Outcomes Assessor
Masking Description: Single-blind (Outcomes Examiner)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (Active Comparator): Soft tissue flap + Connective Tissue Graft
  Interventions: Procedure: Soft tissue flap + Connective Tissue Graft
- Test (Experimental): Soft tissue flap + Geistlich Fibro-Gide®
  Interventions: Device: Soft tissue flap + Geistlich Fibro-Gide®

INTERVENTIONS:
Procedure: Soft tissue flap + Connective Tissue Graft — The treatment site is accessed using a full thickness flap extending at least 1 full tooth mesial and distal, vertical releasing incisions may be used to obtain flap release for full coverage of the treatment site and graft without compression. The harvest graft donor area will be the palate in the bicuspid region on the same side as the control soft tissue augmentation therapy. The CTG will be harvested using full thickness incisions that include the periosteum and will be closed using suture and coating the incision line with a tissue adhesive. No covering stents or packs should be employed. The CTG will be sling sutured in place and the flap secured using a double sling suturing technique.
  Arms: Control
Device: Soft tissue flap + Geistlich Fibro-Gide® — The treatment site is accessed using a full thickness flap extending at least 1 full tooth mesial and distal, vertical releasing incisions may be used to obtain flap release for full coverage of the treatment site and matrix without compression. Geistlich Fibro-Gide® is cut to shape to the treatment site and placed dry into the site. The flap is secured using a double sling suturing technique.
  Arms: Test

SUMMARY:
This double blind, randomized, parallel study evaluates the non-inferiority of Geistlich Fibro-Gide® in comparison to connective tissue graft for soft tissue volume augmentation around dental implants

DETAILED DESCRIPTION:
A total sample size of 60 subjects (n=60) will be evaluated at 5 centers, by 6 Investigators with approximately 10-subjects per Investigator. Power analysis based on 80% power, past Thoma, Zeltner and González-Martin studies 1,2,3 and a one-sided confidence interval of 0.025, indicates that with a volume change standard deviation between 0.5 and 0.7 mm, 17-31 subjects are required per group (test and control), so 50-60 subjects are an acceptable estimate, with a preference for 60, given potential loss to long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects requiring soft tissue augmentation around single implants, i.e., thin biotype with potential for
* All implants must be at least 6 months post bone graft/implant placement
* have at least 1 mm of keratinized tissue width (KTw),
* have final restoration permanently in place for at least 4-weeks and
* subject have no recession on the implant body
* Subjects who, can achieve good oral hygiene (80% plaque free surfaces on the implant and maintain 80% plaque free surfaces on teeth adjacent to treatment sites).

Exclusion Criteria:

* participation within the last six months in other interventional studies.
* any systemic condition that could influence healing, such as uncontrolled diabetes mellitus - confirmed by A1C score ≥7% - cancer, HIV, oral muco- cutaneous conditions and drug induced gingival enlargement.
* taking medications that compromise wound healing, such as chronic steroid use - either inhaler or systemic, calcium channel blockers with secondary hyperplastic tissue reactions, anti-seizure medications, IV bisphosphates for bone metabolic diseases, radiation or other immuno-suppressive therapy.
* acute infectious lesions in the areas intended for surgery.
* History within the last 6 months of weekly or more frequent use of nicotine products
* Female subjects who are pregnant or lactating, or sexually active female subjects who are of childbearing potential and who are not using hormonal or barrier methods of birth control
* Untreated, moderate to severe periodontal disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-13 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in gingival soft tissue volume assessed with 3D scanning | 6 months post treatment
  Change in gingival soft tissue volume compared to baseline [Time Frame 6 months post-treatment] Measured by digital contour scan

SECONDARY OUTCOMES:
All Adverse Events, serious and non serious | Day 0, after 2, 4, 12weeks, 6 Months, 1,3,5 Years
  Recording and Assessment of all (S)AEs starting from Visit 2 onwards, Surgery
Post-OP Patient Reported Outcome Questionnaire | 6 Months, 1,3,5 Years
  subjects will answer a questionnaire regarding discomfort, esthetic satisfaction and overall satisfaction questions asked by a 3rd-party rec
  At Visits 2-weeks, and 1- and 3-months post-operative, subjects will answer discomfort/ pain questions asked by a 3rd-party recorder.
Concomitant medication | 2,4,12 weeks, 6 months, 1,3,5 Years
  Concomitant medication review compared with Visit 1 and 2
Change in gingival soft tissue contour | 3 months, 1,3, 5 Years
  soft tissue contour measured digitally ( 3D-scan) and compared with baseline
General Periodontal Examination (GPE) | 4, 12 weeks, 6 Months, 1,3,5 Years
  Changes of GPE at various visits compared to baseline,
Pink esthetic score (PES) | 6 Months, 1,3,5 Years
  pink esthetic score evaluates soft tissue around single-tooth implants. The PES is based on seven variables: Mesial papilla, Distal papilla, Soft tissue Level, Soft-tissue contour, Alveolar process deficiency, Soft-tissue Color, Soft tissue texture, 2-1-0 score

CONTACTS AND LOCATIONS:
Overall Officials: Donald S Clem III, DDS, Principal Investigator — Regenative Solutions
Locations (5):
- United States (5):
  - Regenerative Solutions, Fullerton, California
  - McClain Schallhorn Periodonitcs, Aurora, Colorado
  - Perio Health Professionals, Houston, Texas
  - Periodontal and Dental Implant Surgical Specialist, Virginia Beach, Virginia
  - Santarelli Oral and Facial Surgery, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No